CLINICAL TRIAL: NCT03835312
Title: Sequential Transplantation of Umbilical Cord Blood Stem Cells and Islet Cells in Children and Adolescents With Monogenic Immunodeficiency Type 1 Diabetes Mellitus
Brief Title: Sequential Transplantation of UCBSCs and Islet Cells in Children and Adolescents With Monogenic Immunodeficiency T1DM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SeqTranUCBC&IC-001
Record Dates: First submitted 2019-01-31; First posted 2019-02-08 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus, Type 1; Immunologic Deficiency Syndromes
Keywords: Islets of Langerhans Transplantation; Cord Blood Stem Cell Transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Immunologic Deficiency Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Sequential transplantation of umbilical cord blood stem cells and islet cells
  Interventions: Procedure: Sequential transplantation

INTERVENTIONS:
Procedure: Sequential transplantation — After successful matching of umbilical cord blood stem cells, patients will receive pretreatment and chemotherapy under protective isolation, followed by thawing and reinfusion of umbilical cord blood stem cells. Immunosuppressive agents will be used for GVHD prevention and anti-infection support will be provided after reinfusion. The status of umbilical cord blood stem cell implantation, immune reconstruction and therapeutic effect will be evaluated. Islet transplantation will be performed in those who meet the conditions. The long-term prognosis will be observed by long-term follow-up.

SUMMARY:
This study evaluates the efficacy of sequential transplantation of umbilical cord blood stem cells and islet cells in children with monogenic immunodeficiency type 1 diabetes mellitus. Umbilical cord blood stem cell transplantation will be performed first. Children with stable immune reconstruction will than receive islet cell transplantation.

DETAILED DESCRIPTION:
Monogenic immunodeficiency type 1 diabetes mellitus (T1DM) usually onsets in early age and has a long course of treatment. Because of T cell deficiency, patients are prone to recurrent infection, hemorrhage, sepsis, colitis or complications of diabetes mellitus, which lead to early death.

New clinical treatment schemes have been explored and introduced around the world. Sequential transplantation of umbilical cord blood stem cells and islet cells is the latest treatment method for these children. Early treatment of monogenic immunodeficiency T1DM children can avoid disease-related organ toxicity, infection risk associated with chronic immunosuppression, and possible prevention of autoimmune endocrine organ damage. Thus, sequential transplantation of umbilical cord blood stem cells and islet cells is the only possible cure for those patients currently.

ELIGIBILITY:
Inclusion Criteria:

1.Type 1 diabetes mellitus children with genetic immunodeficiency

1. Meet the diagnostic criteria of type 1 diabetes mellitus: clinical manifestations of typical diabetes mellitus include polyphagia, polyuria, weight loss, or diabetic ketoacidosis, confirmed by blood sugar level, islet function and autoimmune antibody.
2. Existence of extrapancreatic organ damage: (1) inflammatory bowel disease, (2) impairment of renal function, (3) repeated infection of mouth, skin, anus or whole body, (4) immune hepatitis, (5) persistent chronic immune iridocyclitis, (6) immune adrenalinitis leading to adrenocortical dysfunction, (7) pituitary inflammation leading to hypophysis, (8) rheumatoid disease, (9) immune vasculitis, (10) systemic lupus erythematosus, (11) other organs besides thyroid function damage. Suffering from one or more of above diseases. Recurrence after receiving regular clinical treatment, including symptomatic treatment of organ protective drugs.
3. Gene mutation was found according to gene diagnosis: gene mutation was found by gene sequencing. Literature searches at home and abroad confirmed that the defect of the gene resulted in autoimmune or immune dysfunction, resulting in multiple organ dysfunction and poor prognosis.

Exclusion Criteria:

1. Mature and effective treatment methods are available.
2. HIV, HBV and HCV were positive.
3. A the active period of infection.
4. At the active stage of malignant tumors.
5. Combination of other fatal diseases.
6. Existence of mental and psychological diseases.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of serum C-peptide | from the completion of treatment to 3 months
  Islet function (concentration of serum C-peptide)
Concentration of serum C-peptide | from the completion of treatment to 3 years
  Islet function (concentration of serum C-peptide)

SECONDARY OUTCOMES:
Concentration of serum C-peptide | from the completion of treatment to 6 months
  Islet function (concentration of serum C-peptide)
Concentration of serum C-peptide | from the completion of treatment to 9 months
  Islet function (concentration of serum C-peptide)
Concentration of serum C-peptide | from the completion of treatment to 12 months
  Islet function (concentration of serum C-peptide)
Concentration of serum C-peptide | from the completion of treatment to 15 months
  Islet function (concentration of serum C-peptide)
Concentration of serum C-peptide | from the completion of treatment to 18 months
  Islet function (concentration of serum C-peptide)
Concentration of serum C-peptide | from the completion of treatment to 21 months
  Islet function (concentration of serum C-peptide)
Concentration of serum C-peptide | from the completion of treatment to 24 months
  Islet function (concentration of serum C-peptide)
Concentration of serum C-peptide | from the completion of treatment to 27 months
  Islet function (concentration of serum C-peptide)
Concentration of serum C-peptide | from the completion of treatment to 30 months
  Islet function (concentration of serum C-peptide)
Concentration of serum C-peptide | from the completion of treatment to 33 months
  Islet function (concentration of serum C-peptide)
Concentration of serum insulin | from the completion of treatment to 3 months
  Concentration of serum insulin
Concentration of serum insulin | from the completion of treatment to 6 months
  Concentration of serum insulin
Concentration of serum insulin | from the completion of treatment to 9 months
  Concentration of serum insulin
Concentration of serum insulin | from the completion of treatment to 12 months
  Concentration of serum insulin
Concentration of serum insulin | from the completion of treatment to 15 months
  Concentration of serum insulin
Concentration of serum insulin | from the completion of treatment to 18 months
  Concentration of serum insulin
Concentration of serum insulin | from the completion of treatment to 21 months
  Concentration of serum insulin
Concentration of serum insulin | from the completion of treatment to 24 months
  Concentration of serum insulin
Concentration of serum insulin | from the completion of treatment to 27 months
  Concentration of serum insulin
Concentration of serum insulin | from the completion of treatment to 30 months
  Concentration of serum insulin
Concentration of serum insulin | from the completion of treatment to 33 months
  Concentration of serum insulin
Concentration of serum insulin | from the completion of treatment to 36 months
  Concentration of serum insulin
Fast blood glucose level | from the completion of treatment to 3 months
  Fast blood glucose level
Fast blood glucose level | from the completion of treatment to 6 months
  Fast blood glucose level
Fast blood glucose level | from the completion of treatment to 9 months
  Fast blood glucose level
Fast blood glucose level | from the completion of treatment to 12 months
  Fast blood glucose level
Fast blood glucose level | from the completion of treatment to 15 months
  Fast blood glucose level
Fast blood glucose level | from the completion of treatment to 18 months
  Fast blood glucose level
Fast blood glucose level | from the completion of treatment to 21 months
  Fast blood glucose level
Fast blood glucose level | from the completion of treatment to 24 months
  Fast blood glucose level
Fast blood glucose level | from the completion of treatment to 27 months
  Fast blood glucose level
Fast blood glucose level | from the completion of treatment to 30 months
  Fast blood glucose level
Fast blood glucose level | from the completion of treatment to 33 months
  Fast blood glucose level
Fast blood glucose level | from the completion of treatment to 36 months
  Fast blood glucose level
HbA1c level | from the completion of treatment to 3 months
  HbA1c level
HbA1c level | from the completion of treatment to 6 months
  HbA1c level
HbA1c level | from the completion of treatment to 9 months
  HbA1c level
HbA1c level | from the completion of treatment to 12 months
  HbA1c level
HbA1c level | from the completion of treatment to 15 months
  HbA1c level
HbA1c level | from the completion of treatment to 18 months
  HbA1c level
HbA1c level | from the completion of treatment to 21 months
  HbA1c level
HbA1c level | from the completion of treatment to 24 months
  HbA1c level
HbA1c level | from the completion of treatment to 27 months
  HbA1c level
HbA1c level | from the completion of treatment to 30 months
  HbA1c level
HbA1c level | from the completion of treatment to 33 months
  HbA1c level
HbA1c level | from the completion of treatment to 36 months
  HbA1c level
occurrence of infection (number of infections) | from the completion of treatment to 3 months
  occurrence of infection (number of infections)
occurrence of infection (number of infections) | from the completion of treatment to 6 months
  occurrence of infection (number of infections)
occurrence of infection (number of infections) | from the completion of treatment to 9 months
  occurrence of infection (number of infections)
occurrence of infection (number of infections) | from the completion of treatment to 12 months
  occurrence of infection (number of infections)
occurrence of infection (number of infections) | from the completion of treatment to 15 months
  occurrence of infection (number of infections)
occurrence of infection (number of infections) | from the completion of treatment to 18 months
  occurrence of infection (number of infections)
occurrence of infection (number of infections) | from the completion of treatment to 21 months
  occurrence of infection (number of infections)
occurrence of infection (number of infections) | from the completion of treatment to 24 months
  occurrence of infection (number of infections)
occurrence of infection (number of infections) | from the completion of treatment to 27 months
  occurrence of infection (number of infections)
occurrence of infection (number of infections) | from the completion of treatment to 30 months
  occurrence of infection (number of infections)
occurrence of infection (number of infections) | from the completion of treatment to 33 months
  occurrence of infection (number of infections)
occurrence of infection (number of infections) | from the completion of treatment to 36 months
  occurrence of infection (number of infections)
Concentration of blood immunoglobulin | from the completion of treatment to 3 months
  Concentration of blood immunoglobulin
Concentration of blood immunoglobulin | from the completion of treatment to 6 months
  Concentration of blood immunoglobulin
Concentration of blood immunoglobulin | from the completion of treatment to 9 months
  Concentration of blood immunoglobulin
Concentration of blood immunoglobulin | from the completion of treatment to 12 months
  Concentration of blood immunoglobulin
Concentration of blood immunoglobulin | from the completion of treatment to 15 months
  Concentration of blood immunoglobulin
Concentration of blood immunoglobulin | from the completion of treatment to 18 months
  Concentration of blood immunoglobulin
Concentration of blood immunoglobulin | from the completion of treatment to 21 months
  Concentration of blood immunoglobulin
Concentration of blood immunoglobulin | from the completion of treatment to 24 months
  Concentration of blood immunoglobulin
Concentration of blood immunoglobulin | from the completion of treatment to 27 months
  Concentration of blood immunoglobulin
Concentration of blood immunoglobulin | from the completion of treatment to 30 months
  Concentration of blood immunoglobulin
Concentration of blood immunoglobulin | from the completion of treatment to 33 months
  Concentration of blood immunoglobulin
Concentration of blood immunoglobulin | from the completion of treatment to 36 months
  Concentration of blood immunoglobulin
Concentration of T lymphocyte subsets | from the completion of treatment to 3 months
  Concentration of T lymphocyte subsets
Concentration of T lymphocyte subsets | from the completion of treatment to 6 months
  Concentration of T lymphocyte subsets
Concentration of T lymphocyte subsets | from the completion of treatment to 9 months
  Concentration of T lymphocyte subsets
Concentration of T lymphocyte subsets | from the completion of treatment to 12 months
  Concentration of T lymphocyte subsets
Concentration of T lymphocyte subsets | from the completion of treatment to 15 months
  Concentration of T lymphocyte subsets
Concentration of T lymphocyte subsets | from the completion of treatment to 18 months
  Concentration of T lymphocyte subsets
Concentration of T lymphocyte subsets | from the completion of treatment to 21 months
  Concentration of T lymphocyte subsets
Concentration of T lymphocyte subsets | from the completion of treatment to 24 months
  Concentration of T lymphocyte subsets
Concentration of T lymphocyte subsets | from the completion of treatment to 27 months
  Concentration of T lymphocyte subsets
Concentration of T lymphocyte subsets | from the completion of treatment to 30 months
  Concentration of T lymphocyte subsets
Concentration of T lymphocyte subsets | from the completion of treatment to 33 months
  Concentration of T lymphocyte subsets
Concentration of T lymphocyte subsets | from the completion of treatment to 36 months
  Concentration of T lymphocyte subsets
Concentraion of interleukin-2 | from the completion of treatment to 3 months
  Cytokines (concentraion of interleukin-2)
Concentraion of interleukin-2 | from the completion of treatment to 6 months
  Cytokines (concentraion of interleukin-2)
Concentraion of interleukin-2 | from the completion of treatment to 9 months
  Cytokines (concentraion of interleukin-2)
Concentraion of interleukin-2 | from the completion of treatment to 12 months
  Cytokines (concentraion of interleukin-2)
Concentraion of interleukin-2 | from the completion of treatment to 15 months
  Cytokines (concentraion of interleukin-2)
Concentraion of interleukin-2 | from the completion of treatment to 18 months
  Cytokines (concentraion of interleukin-2)
Concentraion of interleukin-2 | from the completion of treatment to 21 months
  Cytokines (concentraion of interleukin-2)
Concentraion of interleukin-2 | from the completion of treatment to 24 months
  Cytokines (concentraion of interleukin-2)
Concentraion of interleukin-2 | from the completion of treatment to 27 months
  Cytokines (concentraion of interleukin-2)
Concentraion of interleukin-2 | from the completion of treatment to 30 months
  Cytokines (concentraion of interleukin-2)
Concentraion of interleukin-2 | from the completion of treatment to 33 months
  Cytokines (concentraion of interleukin-2)
Concentraion of interleukin-2 | from the completion of treatment to 36 months
  Cytokines (concentraion of interleukin-2)
Body height | from the completion of treatment to 3 months
  Body height
Body height | from the completion of treatment to 6 months
  Body height
Body height | from the completion of treatment to 9 months
  Body height
Body height | from the completion of treatment to 12 months
  Body height
Body height | from the completion of treatment to 15 months
  Body height
Body height | from the completion of treatment to 18 months
  Body height
Body height | from the completion of treatment to 21 months
  Body height
Body height | from the completion of treatment to 24 months
  Body height
Body height | from the completion of treatment to 27 months
  Body height
Body height | from the completion of treatment to 30 months
  Body height
Body height | from the completion of treatment to 33 months
  Body height
Body height | from the completion of treatment to 36 months
  Body height
Body weight | from the completion of treatment to 3 months
  Body weight
Body weight | from the completion of treatment to 6 months
  Body weight
Body weight | from the completion of treatment to 9 months
  Body weight
Body weight | from the completion of treatment to 12 months
  Body weight
Body weight | from the completion of treatment to 15 months
  Body weight
Body weight | from the completion of treatment to 18 months
  Body weight
Body weight | from the completion of treatment to 21 months
  Body weight
Body weight | from the completion of treatment to 24 months
  Body weight
Body weight | from the completion of treatment to 27 months
  Body weight
Body weight | from the completion of treatment to 30 months
  Body weight
Body weight | from the completion of treatment to 33 months
  Body weight
Body weight | from the completion of treatment to 36 months
  Body weight
Tanner stage | from the completion of treatment to 3 months
  Puberty change (Tanner stage)
Tanner stage | from the completion of treatment to 6 months
  Puberty change (Tanner stage)
Tanner stage | from the completion of treatment to 9 months
  Puberty change (Tanner stage)
Tanner stage | from the completion of treatment to 12 months
  Puberty change (Tanner stage)
Tanner stage | from the completion of treatment to 15 months
  Puberty change (Tanner stage)
Tanner stage | from the completion of treatment to 18 months
  Puberty change (Tanner stage)
Tanner stage | from the completion of treatment to 21 months
  Puberty change (Tanner stage)
Tanner stage | from the completion of treatment to 24 months
  Puberty change (Tanner stage)
Tanner stage | from the completion of treatment to 27 months
  Puberty change (Tanner stage)
Tanner stage | from the completion of treatment to 30 months
  Puberty change (Tanner stage)
Tanner stage | from the completion of treatment to 33 months
  Puberty change (Tanner stage)
Tanner stage | from the completion of treatment to 36 months
  Puberty change (Tanner stage)
Occurrence of graft versus host disease | from the completion of treatment to 3 months
  Occurrence of graft versus host disease
Occurrence of graft versus host disease | from the completion of treatment to 6 months
  Occurrence of graft versus host disease
Occurrence of graft versus host disease | from the completion of treatment to 9 months
  Occurrence of graft versus host disease
Occurrence of graft versus host disease | from the completion of treatment to 12 months
  Occurrence of graft versus host disease
Occurrence of graft versus host disease | from the completion of treatment to 15 months
  Occurrence of graft versus host disease
Occurrence of graft versus host disease | from the completion of treatment to 18 months
  Occurrence of graft versus host disease
Occurrence of graft versus host disease | from the completion of treatment to 21 months
  Occurrence of graft versus host disease
Occurrence of graft versus host disease | from the completion of treatment to 24 months
  Occurrence of graft versus host disease
Occurrence of graft versus host disease | from the completion of treatment to 27 months
  Occurrence of graft versus host disease
Occurrence of graft versus host disease | from the completion of treatment to 30 months
  Occurrence of graft versus host disease
Occurrence of graft versus host disease | from the completion of treatment to 33 months
  Occurrence of graft versus host disease
Occurrence of graft versus host disease | from the completion of treatment to 36 months
  Occurrence of graft versus host disease

CONTACTS AND LOCATIONS:
Overall Officials: Luo Feihong, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho NH, Shaw JE, Karuranga S, Huang Y, da Rocha Fernandes JD, Ohlrogge AW, Malanda B. IDF Diabetes Atlas: Global estimates of diabetes prevalence for 2017 and projections for 2045. Diabetes Res Clin Pract. 2018 Apr;138:271-281. doi: 10.1016/j.diabres.2018.02.023. Epub 2018 Feb 26. PMID 29496507
- [Background] Fu H, Shen SX, Chen ZW, Wang JJ, Ye TT, LaPorte RE, Tajima N. Shanghai, China, has the lowest confirmed incidence of childhood diabetes in the world. Diabetes Care. 1994 Oct;17(10):1206-8. doi: 10.2337/diacare.17.10.1206. PMID 7821146
- [Background] Zhao Z, Sun C, Wang C, Li P, Wang W, Ye J, Gu X, Wang X, Shen S, Zhi D, Lu Z, Ye R, Cheng R, Xi L, Li X, Zheng Z, Zhang M, Luo F. Rapidly rising incidence of childhood type 1 diabetes in Chinese population: epidemiology in Shanghai during 1997-2011. Acta Diabetol. 2014 Dec;51(6):947-53. doi: 10.1007/s00592-014-0590-2. Epub 2014 Apr 29. PMID 24777734
- [Background] Daniels M, DuBose SN, Maahs DM, Beck RW, Fox LA, Gubitosi-Klug R, Laffel LM, Miller KM, Speer H, Tamborlane WV, Tansey MJ; T1D Exchange Clinic Network. Factors associated with microalbuminuria in 7,549 children and adolescents with type 1 diabetes in the T1D Exchange clinic registry. Diabetes Care. 2013 Sep;36(9):2639-45. doi: 10.2337/dc12-2192. Epub 2013 Apr 22. PMID 23610082
- [Background] Amin R, Widmer B, Prevost AT, Schwarze P, Cooper J, Edge J, Marcovecchio L, Neil A, Dalton RN, Dunger DB. Risk of microalbuminuria and progression to macroalbuminuria in a cohort with childhood onset type 1 diabetes: prospective observational study. BMJ. 2008 Mar 29;336(7646):697-701. doi: 10.1136/bmj.39478.378241.BE. Epub 2008 Mar 18. PMID 18349042
- [Background] Mollsten A, Svensson M, Waernbaum I, Berhan Y, Schon S, Nystrom L, Arnqvist HJ, Dahlquist G; Swedish Childhood Diabetes Study Group; Diabetes Incidence Study in Sweden; Swedish Renal Registry. Cumulative risk, age at onset, and sex-specific differences for developing end-stage renal disease in young patients with type 1 diabetes: a nationwide population-based cohort study. Diabetes. 2010 Jul;59(7):1803-8. doi: 10.2337/db09-1744. Epub 2010 Apr 27. PMID 20424230
- [Background] American Diabetes Association. (2) Classification and diagnosis of diabetes. Diabetes Care. 2015 Jan;38 Suppl:S8-S16. doi: 10.2337/dc15-S005. No abstract available. PMID 25537714
- [Background] Wildin RS, Smyk-Pearson S, Filipovich AH. Clinical and molecular features of the immunodysregulation, polyendocrinopathy, enteropathy, X linked (IPEX) syndrome. J Med Genet. 2002 Aug;39(8):537-45. doi: 10.1136/jmg.39.8.537. PMID 12161590
- [Background] Uzel G, Sampaio EP, Lawrence MG, Hsu AP, Hackett M, Dorsey MJ, Noel RJ, Verbsky JW, Freeman AF, Janssen E, Bonilla FA, Pechacek J, Chandrasekaran P, Browne SK, Agharahimi A, Gharib AM, Mannurita SC, Yim JJ, Gambineri E, Torgerson T, Tran DQ, Milner JD, Holland SM. Dominant gain-of-function STAT1 mutations in FOXP3 wild-type immune dysregulation-polyendocrinopathy-enteropathy-X-linked-like syndrome. J Allergy Clin Immunol. 2013 Jun;131(6):1611-23. doi: 10.1016/j.jaci.2012.11.054. Epub 2013 Mar 25. PMID 23534974
- [Background] Bennett CL, Christie J, Ramsdell F, Brunkow ME, Ferguson PJ, Whitesell L, Kelly TE, Saulsbury FT, Chance PF, Ochs HD. The immune dysregulation, polyendocrinopathy, enteropathy, X-linked syndrome (IPEX) is caused by mutations of FOXP3. Nat Genet. 2001 Jan;27(1):20-1. doi: 10.1038/83713. PMID 11137993
- [Background] Rao A, Kamani N, Filipovich A, Lee SM, Davies SM, Dalal J, Shenoy S. Successful bone marrow transplantation for IPEX syndrome after reduced-intensity conditioning. Blood. 2007 Jan 1;109(1):383-5. doi: 10.1182/blood-2006-05-025072. Epub 2006 Sep 21. PMID 16990602
- [Background] van de Veerdonk FL, Plantinga TS, Hoischen A, Smeekens SP, Joosten LA, Gilissen C, Arts P, Rosentul DC, Carmichael AJ, Smits-van der Graaf CA, Kullberg BJ, van der Meer JW, Lilic D, Veltman JA, Netea MG. STAT1 mutations in autosomal dominant chronic mucocutaneous candidiasis. N Engl J Med. 2011 Jul 7;365(1):54-61. doi: 10.1056/NEJMoa1100102. Epub 2011 Jun 29. PMID 21714643
- [Background] Toubiana J, Okada S, Hiller J, Oleastro M, Lagos Gomez M, Aldave Becerra JC, Ouachee-Chardin M, Fouyssac F, Girisha KM, Etzioni A, Van Montfrans J, Camcioglu Y, Kerns LA, Belohradsky B, Blanche S, Bousfiha A, Rodriguez-Gallego C, Meyts I, Kisand K, Reichenbach J, Renner ED, Rosenzweig S, Grimbacher B, van de Veerdonk FL, Traidl-Hoffmann C, Picard C, Marodi L, Morio T, Kobayashi M, Lilic D, Milner JD, Holland S, Casanova JL, Puel A; International STAT1 Gain-of-Function Study Group. Heterozygous STAT1 gain-of-function mutations underlie an unexpectedly broad clinical phenotype. Blood. 2016 Jun 23;127(25):3154-64. doi: 10.1182/blood-2015-11-679902. Epub 2016 Apr 25. PMID 27114460
- [Background] Leiding JW, Okada S, Hagin D, Abinun M, Shcherbina A, Balashov DN, Kim VHD, Ovadia A, Guthery SL, Pulsipher M, Lilic D, Devlin LA, Christie S, Depner M, Fuchs S, van Royen-Kerkhof A, Lindemans C, Petrovic A, Sullivan KE, Bunin N, Kilic SS, Arpaci F, Calle-Martin O, Martinez-Martinez L, Aldave JC, Kobayashi M, Ohkawa T, Imai K, Iguchi A, Roifman CM, Gennery AR, Slatter M, Ochs HD, Morio T, Torgerson TR; Inborn Errors Working Party of the European Society for Blood and Marrow Transplantation and the Primary Immune Deficiency Treatment Consortium. Hematopoietic stem cell transplantation in patients with gain-of-function signal transducer and activator of transcription 1 mutations. J Allergy Clin Immunol. 2018 Feb;141(2):704-717.e5. doi: 10.1016/j.jaci.2017.03.049. Epub 2017 Jun 7. PMID 28601685
- [Background] Niclauss N, Morel P, Berney T. Has the gap between pancreas and islet transplantation closed? Transplantation. 2014 Sep 27;98(6):593-9. doi: 10.1097/TP.0000000000000288. PMID 25029387
- [Background] Ahearn AJ, Parekh JR, Posselt AM. Islet transplantation for Type 1 diabetes: where are we now? Expert Rev Clin Immunol. 2015 Jan;11(1):59-68. doi: 10.1586/1744666X.2015.978291. Epub 2014 Dec 2. PMID 25454816
- [Background] Kopan C, Tucker T, Alexander M, Mohammadi MR, Pone EJ, Lakey JRT. Approaches in Immunotherapy, Regenerative Medicine, and Bioengineering for Type 1 Diabetes. Front Immunol. 2018 Jun 12;9:1354. doi: 10.3389/fimmu.2018.01354. eCollection 2018. PMID 29963051

DOCUMENTS (3):
  • Study Protocol (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/12/NCT03835312/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/12/NCT03835312/SAP_002.pdf
  • Informed Consent Form (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/12/NCT03835312/ICF_001.pdf